CLINICAL TRIAL: NCT03162744
Title: Methodical Search of Protective Factors During Interview of Suicidal Elderly Patients: Effect on the Proposed Care
Brief Title: Protective Factors Against Elderly Suicide
Acronym: ProFAES
Status: Terminated | Type: Observational
Why Stopped: Inclusion difficulties, Investigator lack of time for the study completion
Sponsor: Groupe Hospitalier de la Rochelle Ré Aunis (Other)
Responsible Party: Sponsor
Other Study IDs: 2015/P08/079
Record Dates: First submitted 2017-05-19; First posted 2017-05-22 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Suicide, Attempted; Suicide Gesture
MeSH Terms: conditions — Suicide, Attempted

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Suicide attempt or ideas: Elderly patients who attempted suicide or who emitted suicidal ideas
  Interventions: Behavioral: Post-suicidal crisis interview

INTERVENTIONS:
Behavioral: Post-suicidal crisis interview — Protective factor exploration during post-suicidal crisis interview

SUMMARY:
Suicidal intentionality is generally stronger among the elderly, suicidal acts are more violent and are combined with a greater physical fragility. The suicide of an older adult is a situation that often leads to helplessness feelings.

Analysis of the literature reveals two types of major interventions in order to reduce suicide rate: reducing risk factors and increasing protective factors. Risk factors are well documented, particularly from studies using psychological autopsies. However, protective factors are much less studied for the elderly. Yet the identification of relevant and available protective mechanisms in a suicidal crisis is essential to effectively guide nurses and health professionals in therapeutic commitment and intervention.

DETAILED DESCRIPTION:
France has a suicide rate (16.2 per 100 000 inhabitants) well above the European average rate (10.2 per 100 000 inhabitants). The Poitou-Charentes region is in a situation of excess mortality by suicide compared to France (+ 25%). While the ratio of suicide attempts per suicide is about 200/1 before 25 years, it is estimated to be 4/1 after 65 years, or even 1/1 in elderly men. In France, suicide attempts are not systematically recorded and the frequency of suicidal ideation is poorly understood. The consensus conference on suicidal crisis highlights a number of clinical points specific to the elderly population (suicidal ideas are not always clearly expressed or unidentified, there are various manifestations of the psychic crisis, greater vulnerability of this population), but the complexity of interactions between suicidal risk factors limits our predictive capabilities of suicidal intention in an elderly person. Analysis of the literature reveals two types of major interventions in order to reduce the suicide rate: those aimed at reducing risk factors and those aimed at increasing protective factors. The objective of our research is to determine the effect of protective factor methodical search on post-crisis patient care.

ELIGIBILITY:
Inclusion Criteria:

* Attempted suicide and / or suicidal ideas
* Informed and agreed to participate

Exclusion Criteria:

* Cognitive disorders
* Refusal to participate

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients will be screened in the psychiatric, geriatric and emergency departments of la Rochelle and Rochefort secondary hospitals
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2018-02-16 (Actual); Primary Completion 2019-02-16 (Actual); Study Completion 2019-05-27 (Actual)

PRIMARY OUTCOMES:
Number of outpatients (with a low to moderate risk of suicidal recurrence) | 7 days
  Based on risk, emergency and hazard, patients are classified as being at low, moderate and high risk of suicidal recurrence. Patients with low to moderate risk of suicidal recurrence are either inpatient or outpatient.

SECONDARY OUTCOMES:
Number of patients considering themselves to be in good health | 7 days
  Score > 0 at Health Status questionnaire (SF36) item 1
Number of patients considering that their physical or mental state did not alter their social life | 7 days
  Score > 50 at Health Status questionnaire (SF36) items 6 or 10
Number of patients maintaining autonomy | 7 days
  Score = 0 at Instrumental Activities of Daily Living scale
Number of patients with religious practice | 7 days
  Binary answer from patients (yes/no I have a religious practice)
Number of patients with a sense of success and self-esteem | 7 days
  Binary answer from patients (yes/no I have a a sense of success and self-esteem)
Number of patients considering their family environment to be satisfactory | 7 days
  Binary answer from patients (yes/no I am satisfied with my family environment)
Number of patients with at least one environmental protection factor | 7 days
  Friendly network, associative investment, volunteering, specialized care, recreation, positive image from the entourage, presence of a third party, housekeeper, postman, pet, shopping facilities, doctor, pharmacy ...
Number of patients with social protection factors | 7 days
  Easy access to Health facilities, sufficient financial income
Number of patients able to adapt to difficult situations | 7 days
  score ≤ 12 at Neo Personality Inventory vulnerability item
Number of patients with extraversion capabilities | 7 days
  score ≥ 20 at Neo Personality Inventory extraversion item
Number of patients with openness to others | 7 days
  score ≥ 20 at Neo Personality Inventory Openness to feelings item
Number of patients considering that their health has improved | 3 months
  Patients will be asked if they feel that their health has improved, has not changed or has worsened

CONTACTS AND LOCATIONS:
Overall Officials: Karine REISS, MD, Study Director — Groupe Hospitalier de la Rochelle Ré Aunis
Locations (1):
- Groupe Hospitalier de la Rochelle Ré Aunis, La Rochelle, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Richard-Devantoy S, Jollant F. [Suicide in the elderly: age-related specificities?]. Sante Ment Que. 2012 Autumn;37(2):151-73. doi: 10.7202/1014949ar. French. PMID 23666286
- [Background] Conwell Y, Thompson C. Suicidal behavior in elders. Psychiatr Clin North Am. 2008 Jun;31(2):333-56. doi: 10.1016/j.psc.2008.01.004. PMID 18439452
- [Background] Casadebaig F, Ruffin D, Philippe A. [Suicide in the elderly at home and in retirement homes in France]. Rev Epidemiol Sante Publique. 2003 Feb;51(1 Pt 1):55-64. French. PMID 12684581
- See also: Epidemiology of suicide in France — https://www.insee.fr/fr/statistiques